CLINICAL TRIAL: NCT00875030
Title: A Single-Dose Bioequivalence Study Comparing Artesunate Sachets (Pfizer) To Arsuamoon® Tablets (Guilin-China) In Healthy Subjects
Brief Title: A Study Comparing Blood Levels After Single-Dose Administration Of Artesunate Sachets (Pfizer) Versus Single-Dose Administration Of Arsuamoon® Tablets (Guilin-China) In Healthy Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: B0551002
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Last update posted 2010-06-09 (Estimated); Status verified 2010-06

CONDITIONS: Healthy Volunteers
Keywords: Bioequivalence study-artesunate sachets-arsuamoon tablet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1.0 (Experimental)
  Interventions: Drug: artesunate sachets
- 2.0 (Active Comparator)
  Interventions: Drug: Arsuamoon

INTERVENTIONS:
Drug: artesunate sachets — single dose 50 mg (2 X 25 mg) artesunate sachets
  Arms: 1.0
Drug: Arsuamoon — single dose 50 mg arsuamoon tablet
  Arms: 2.0

SUMMARY:
The primary objective of the study is to determine bioequivalence of 50 mg (2x25 mg) Artesunate Sachet (Pfizer) versus 50 mg (1x50 mg) tablet, Arsuamoon® (Guilin China) which is the World Health Organization Reference standard for artesunate The secondary objective is to assess the safety of Artesunate Sachet (Pfizer) and Arsuamoon® tablet (Guilin China).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years, inclusive.
* Body Mass Index (BMI) of 18 to 30 kg/m2; and a total body weight >45 kg (99 lbs).
* An informed consent document signed and dated by the subject or a legally acceptable representative.

Exclusion Criteria:

* Any condition possibly affecting drug absorption.
* A positive urine drug screen.
* Have a known history of hypersensitivity, allergy (except for untreated, asymptomatic, seasonal allergies at the time of dosing), severe adverse drug reaction, or intolerance to artesunate or its derivatives.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2009-06; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Cmax, AUCinf and AUClast, for DHA | 1 year

SECONDARY OUTCOMES:
Tmax and t1/2 for DHA; Cmax, AUCinf, AUClast, Tmax and t1/2 for artesunate. | 1 year
Safety laboratory tests, vital signs, and adverse events. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Navi Mumbai, Maharashtra, India

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0551002&StudyName=A%20Study%20Comparing%20Blood%20Levels%20After%20Single-Dose%20Administration%20Of%20Artesunate%20Sachets%20%28Pfizer%29%20Versus%20Single-Dose%20Administration%20Of%20Arsuam